CLINICAL TRIAL: NCT06225388
Title: Effect of Wearing a Compression Sock During Running on Delayed Onset Muscle Soreness in Distance Runners: A Randomised, Double-blind, Sham-controlled, Crossover Trial.
Brief Title: Effect of Wearing a Compression Sock During Running on Muscle Soreness in Distance Runners.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Gustavo Telles, Principal Investigator, Centro Universitário Augusto Motta
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Muscle Soreness; Perceived Recovery; Perceived Exertion; Affective Response; Heart Rate
Keywords: runner; garments; pain; stocking; knee; sports
MeSH Terms: conditions — Myalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression socks (Experimental): For the intervention, compression socks will be used, composed of 81% polyamide, 15% elastane and 4% polypropylene (Kendall sports, Kendall, São Paulo, Brazil). The sock offers compression of 20 to 30 mmHg in a decreasing manner with greater pressure at the ankle and less pressure at the knee joint line. Based on the manufacturer's guidelines, the sock size will be determined by measuring the calf and ankle circumference.
  Interventions: Other: Compression socks
- Placebo socks (Placebo Comparator): The placebo sock will be represented by a commercial sock composed of 70% polyamide, 24% cotton and 5% elastodiene without the purpose of providing compression.
  Interventions: Other: Placebo socks

INTERVENTIONS:
Other: Compression socks — A pair of socks corresponding to the intervention allocated will be given to the participant, by an investigator who will not participate in the evaluation, in a dark plastic bag to avoid any visual influence. We will adopt strategies to prevent information about the socks from influencing the participants' behaviour: (1) the compression and placebo socks will have the same colour, any visual detail and branding will be covered. Words or logos from the compression sock will be covered, so participants are unable to differentiate them. (2) After performing the running protocol, participants will remove their socks and return them to the investigator.
  Arms: Compression socks
Other: Placebo socks — The compression and placebo socks will have the same colour, any visual detail and branding will be covered. Words or logos from the compression sock will be covered, so participants are unable to differentiate them. (2) After performing the running protocol, participants will remove their socks and return them to the investigator.
  Arms: Placebo socks

SUMMARY:
Running is the most popular physical activity worldwide. Although running provides many health benefits, it is often associated with injuries and symptoms such as delayed onset muscle soreness. There is still a paucity of interventions that can effectively minimise these symptoms in distance runners.

DETAILED DESCRIPTION:
Our primary aim is to explore the effect of compression socks during running on delayed onset muscle soreness after running. Our secondary aims are to explore the effects of compression socks during running on perceived recovery, perceived exertion, affective response, and heart rate after running. This is a randomised, double-blind, sham-controlled crossover trial. Forty-four participants will be recruited via social media, running clubs and the running coaches' network of the research team. Participants will be randomised to complete a running protocol under two conditions (compression socks or sham socks). After that, there will be a wash-out period of 7 to 10 days, and participants will repeat the running protocol under the other conditions. Primary outcome: lower limb muscle soreness will be collected, using a 0-100 numerical pain scale, immediately, 24 hours and 48 hours after the running protocol, with 24 hours post-protocol being the primary timepoint. Secondary outcomes: perceived recovery will be collected, using a 0-10 scale immediately, 24 hours and 48 hours after the running protocol. Perceived exertion, affective response, and heart rate will be registered only immediately after the protocol. Between-group differences will be explored using linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Run consistently in the last six months (at least three times a week and at least 10 kilometres per week);
* Runners who did not run further than 42 kilometres in the last month.

Exclusion Criteria:

* Pregnancy;
* Any lower limbs fracture in the last 12 months;
* History of lower limb arthroplasty or osteotomy, previous venous thrombosis, kidney disease;
* Any running-related injury in the last six months. A running-related injury will be considered the presence of lower limb pain that caused restriction, stoppage of running (distance, speed, duration, or training) for at least seven days or three consecutive scheduled training sessions or the need for a health professional treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Lower limb muscle soreness. | 24 hours post-intervention.
  A visual analogue scale (VAS) will be used to measure the intensity of muscle soreness. This scale ranges from 0 (no pain) to 100 (worst possible pain).

SECONDARY OUTCOMES:
Lower limb muscle soreness. | 5 minutes post-intervention, and 48 hours post-intervention.
  A visual analogue scale (VAS) will be used to measure the intensity of muscle soreness. This scale ranges from 0 (no pain) to 100 (worst possible pain).
Perceived recovery. | 5 minutes post-intervention, 24 hours, and 48 hours post-intervention.
  The Perceived Recovery Status Scales will assess participants' perceived recovery. This scale ranges from 0 (very poorly recovered / extremely tired) to 10 (very well recovered / highly energetic). Values from 0 to 2 indicate "expect declined performance", values from 4 to 6 indicate "expect similar performance", and values from 8 to 10 represent "expect improved performance". Values 3 and 7 are considered transitional conditions. The value 3 means that it is not clear that the participants will be able to maintain their performance, and the value 7 means the participants are not fully recovered
Perceived exertion | 5 minutes post-intervention.
  The Borg Rating of Perceived Exertion (Borg RPE 6-20) will be used assess how hard and strenuous the running protocol was. This scale ranges from 6 (no exertion at all) to 20 (maximal exertion).
Affective response | 5 minutes post-intervention.
  The Feeling Scale is a bipolar scale that measures the affective response (pleasure/displeasure) related to exercise. This scale ranges from + 5 (very good) to - 5 (very bad). Zero is considered neutral; positive values represent pleasure, and negative values represent displeasure.
Heart rate | Through the intervention, an average of 30 minutes.
  The average heart rate in beats per minute will be monitored through a smartwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro AC Nogueira, PhD, Study Chair — Centro Universitário Augusto Motta
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The author will share the study's statistical analysis plan.
Supporting Information: SAP
Access Criteria: The statistical analysis plan will be available upon request.